CLINICAL TRIAL: NCT07203001
Title: An Open-label Phase II Trial to Evaluate the Clinical Efficacy, Safety and Tolerability of MAS825 in Pediatric and Adult Participants With Still's Disease
Brief Title: A Phase II Trial to Evaluate the Clinical Efficacy, Safety and Tolerability of MAS825 in Pediatric and Adult Participants With Still's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMAS825J12201; 2024-520208-25 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2025-09-09; First posted 2025-10-02 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Still´s Disease
Keywords: Still´s disease; pediatric; adult; JIA; AOSD; Juvenile Idiopathic Arthritis; Adult Onset Still s disease; rheumatology; MAS825
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MAS825 (Experimental): Experimental drug
  Interventions: Drug: MAS825

INTERVENTIONS:
Drug: MAS825 — Experimental drug

SUMMARY:
The study is a phase II trial designed to evaluate the clinical efficacy, safety, and tolerability of MAS825 in pediatric and adult participants with Still's disease

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1 with a diagnosis of Still's Disease
* Active diseases defined as:
* CRP or ferritin levels greater than ULN, and any of:

  * Fever ≥ 38°C attributed to Still's Disease activity and documented for a number of days prior to Day 1 or
  * Rash attributed to Still's Disease activity or
  * Musculoskeletal involvement: arthritis in a number of joints per ACP criteria for active joint or
  * Serositis or
  * Macrophage activation syndrome activity as defined by ferritin levels and at least one of: platelet count, a biomarker or fibrinogen levels attributed to Still's Disease activity by the investigator
* Need for glucocorticoids (prednisone or equivalent)

Exclusion Criteria:

* Patients out of weight range
* Ongoing or previous treatment with immunomodulatory drugs

  * A limited number of Still's Disease patients that have previously received MAS825 through a managed access program are permitted on the study
* Glucocorticoid dose exceeding a set limit
* Any conditions or significant medical problems which places the patient at unacceptable risk for MAS825 therapy

  * Still's disease patients with evidence of macrophage activation syndrome are permitted in the study
  * Still's Disease patients with evidence of interstitial lung disease including those requiring supplemental oxygen therapy are permitted in the study
* History of ongoing, chronic or possibly recurrent infection (e.g. HIV, TB, HCV, HBV) and/or symptoms and signs of clinically significant active bacterial, fungal or viral infections
* Live vaccinations within a set time prior to MAS825 treatment. Live vaccines are prohibited up to several months following the last dose
* History of malignancy of any organ system, including post-transplant lymphoproliferative disorder, treated or untreated, within a number of years, regardless of whether there is evidence of local recurrence and metastases
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes or to any of the excipients
* Pregnant or breastfeeding women
* Women of child-bearing potential who do not agree to comply with required contraceptive use

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2029-05-24 (Estimated); Study Completion 2029-05-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinical response based on one set of response criteria | Day 85
  Established measure for efficacy of treatments in the rheumatologic conditions taking into account self-assessment, function and survival.

SECONDARY OUTCOMES:
Number of participants with clinical response based on another set of response criteria | Day 85
  Established measure for efficacy of treatments in the rheumatologic conditions taking into account self-assessment, function and survival.
Response based on a biomarker level | Baseline, Day 85
  To evaluate the efficacy of MAS825 in reducing clinical disease activity
Change in physician assessment based on laboratory features of MAS825 | Baseline, 15 months
  To assess the effect of MAS825 on macrophage activation syndrome
Change from baseline in Glucocorticoid (GC) dose | Baseline, Day 85, Month 6, Month 12
  To evaluate the efficacy of MAS825 as a glucocorticoid-sparing agent
Change from baseline in patient/parent assessment of physical function as assessed by Quality of Life instrument | Baseline, Day 85
  To evaluate the efficacy of MAS825 in improving participant's quality of life
Clinically inactive disease whilst on non-treatment dose corticosteroid at any time during the study | 15 months
  The number of participants with inactive disease will be assessed. Disease activity will be evaluated by the investigator based on physical examination and laboratory parameters.
  Inactive disease is defined according to protocol-specific criteria, which include clinical signs, laboratory values, and physician assessment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Legacy Emanuel Research Hosp Portland, Portland, Oregon
- Novartis Investigative Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.